CLINICAL TRIAL: NCT00955006
Title: A Phase 1b Clinical Trial to Evaluate Mucosal Immune Responses to a DNA Plasmid Vaccine Prime Followed by an HIV-1 Adenoviral Vector Boost in Healthy Adenovirus Type 5 Seronegative HIV-1-uninfected Adults
Brief Title: Immune Response to an HIV DNA Plasmid Vaccine Prime Followed by Adenovirus Boost in HIV-uninfected Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 076; 10625 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

ARMS (1):
- Group 1 (Experimental): Participants will receive three injections of VRC-HIVDNA-016-00-VP at Months, 0, 1, and 2 and one injection of VRCHIVADV014-00-VP at Month 6.
  Interventions: Biological: VRC-HIVDNA-016-00-VP; Biological: VRCHIVADV014-00-VP

INTERVENTIONS:
Biological: VRC-HIVDNA-016-00-VP — Composed of six DNA plasmids in equal concentrations that encode Gag, Pol, and Nef from clade B (strains HXB2, NL4-3, NY5/BRU) and the HIV-1 Env glycoproteins from clade A (strain 92rw020), clade B (strains HXB2/BaL), and clade C (strain 97ZA012). Vaccine will be administered intramuscularly (IM) in the deltoid via needle-free Biojector.
Biological: VRCHIVADV014-00-VP — A mixture of 4 recombinant serotype 5 adenoviral replication deficient vectors, each expressing HIV-1 proteins (clade B Gag-Pol fusion, clade A Env, clade B Env, clade C Env). Administered IM via needle and syringe.

SUMMARY:
The purpose of the study is to determine the safety of mucosal immune responses to a DNA HIV vaccine followed by an adenoviral vector HIV vaccine in HIV uninfected adults.

DETAILED DESCRIPTION:
The worldwide HIV/AIDS epidemic may only be controlled through development of a safe and effective vaccine that will prevent HIV infection. DNA vaccines are inexpensive to construct, readily produced in large quantities, and stable for long periods of time. This study will evaluate the safety and immunogenicity of an experimental multiclade HIV vaccine, VRC-HIVDNA016-00-VP, followed by a similarly structured adenovirus-vectored vaccine boost, VRC-HIVADV014-00-VP, in HIV uninfected adults. The DNA plasmids in both the vaccines code for proteins from HIV subtypes A, B, and C, which together represent 90% of new HIV infections in the world. The study's primary objective is to investigate the ability of a 6-plasmid DNA prime followed by a rAd5 boost to elicit HIV-specific cellular immune responses at mucosal surfaces.

This study will last 12 months and participants will visit the clinic 15 times. Participants will receive three injections of the VRC-HIVDNA016-00-VP vaccine at Months 0, 1, and 2 followed by an injection of VRC-HIVADV014-00-VP at Month 6. All injections will be given in the upper arm. At study visits participants will have a physical, medical history taken, blood collection, and risk reduction counseling. At some visits, rectal biopsies (via anoscopy or, optionally, by flexible sigmoidoscopy), saliva, semen, cervical and/or vaginal fluid samples will also be collected. Pregnancy testing for women will be done prior to each vaccination and study procedure.

Participants will be contacted by study staff once a year for 5 years after the initial study visit for follow-up health and safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Access to participating HVTN CRS and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: participant demonstrates understanding of this study and the Step Study results; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks, amenable to HIV risk reduction counseling, committed to maintaining behavior consistent with low risk of HIV exposure through the last required clinic visit, and willing to continue annual follow-up contact after the last required clinic visit, for a total of 5 years following enrollment
* Agrees not to enroll in another study of an investigational research agent prior to completion of last required protocol clinic visit (excludes annual follow-up contact for safety surveillance)
* Assessed by clinic staff as being at "low risk" for HIV infection. More information on this criterion can be found in the protocol.
* Good general health as shown by medical history, physical exam, and screening laboratory tests. More information on this criterion can be found in the protocol.
* Neutralizing antibody titers of Ad5 less than 1:18
* Hemoglobin equal to or greater than 11.0 g/dL for participants who were born female, 12.5 g/dL for participants who were born male
* White blood cell (WBC) count = 3,300 to 12,000 cells/mm^3
* Total lymphocyte count equal to or greater than 800 cells/mm^3
* Remaining differential either within institutional normal range or accompanied by site physician approval
* Platelets = 125,000 to 550,000/mm^3
* Prothrombin time (PT) less than 1.5 and partial thromboplastin time (PTT) less than 1.25 greater than upper limits of normal
* Alanine transaminase (ALT) is less than 2.5 times the institutional upper limit of normal
* Negative HIV-1 and 2 blood test: participants must have a negative FDA-approved enzyme immunoassay (EIA)
* For participants born female, normal Pap smear or ASCUS with no evidence of high risk HPV within 3 years prior to enrollment
* Participants who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed on the day of initial vaccination prior to vaccination
* Participants who were born female must agree to consistently use effective contraception from at least 21 days prior to enrollment through the last required clinic visit for sexual activity that could lead to pregnancy; or not be of reproductive potential; or be sexually abstinent. More information on this criterion can be found in the protocol.
* Participants who were born female must also agree not to seek pregnancy through alternative methods such as artificial insemination or in vitro fertilization until after the last required clinic visit
* If born male, must be fully circumcised (as documented at a screening examination)

Exclusion Criteria:

* Excessive daily alcohol use or frequent binge drinking or chronic marijuana abuse or any other use of illicit drugs within the past 12 months
* A history of newly acquired syphilis, gonorrhea, non-gonococcal urethritis, herpes simplex virus type 2 (HSV2), Chlamydia, pelvic inflammatory disease (PID), trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B in the past 12 months
* HIV vaccine(s) received in a prior HIV vaccine trial. For potential participants who have received control/placebo in an HIV vaccine trial, the HVTN 076 PSRT will determine eligibility on a case-by-case basis.
* Experimental vaccine(s) received within the last 5 years in a prior vaccine trial. More information on this criterion can be found in the protocol.
* Immunosuppressive medications received within 168 days before first vaccination (eg, oral/parenteral corticosteroids, and/or cytotoxic medications). People taking corticosteroid nasal spray for allergic rhinitis and topical corticosteroids for mild, uncomplicated dermatitis are not excluded.
* Abnormality of the colorectal mucosa, or significant colorectal symptom(s), which in the opinion of the clinician represents a contraindication to biopsy (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa, and presence of hemorrhoids)
* Blood products received within 120 days before first vaccination
* Immunoglobulin received within 60 days before first vaccination
* Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 14 days after vaccination (e.g., measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Influenza vaccine or any vaccines that are not live attenuated vaccines received within 14 days prior to first vaccination or scheduled within 14 days after vaccination (e.g., influenza, tetanus, pneumococcal, hepatitis A or B)
* Investigational research agents received within 30 days before first vaccination
* Intent to participate in another study of an investigational research agent during the planned duration of the study
* Allergy treatment with antigen injections within 30 days before first vaccination or scheduled within 14 days after injection
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. More information on this criterion can be found in the protocol.
* Any medical, psychiatric, or social condition, or occupational or other responsibility that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent
* Serious adverse reactions to vaccines including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. Participants who had a nonanaphylactic adverse reaction to pertussis vaccine as a child are not excluded.
* Autoimmune disease
* Immunodeficiency
* Active syphilis infection. (Not excluded: syphilis fully treated over 6 months prior to enrollment)
* Reports one or more perianal HSV outbreaks within 30 days prior to enrollment
* Positive gonorrhea or Chlamydia urine nucleic acid amplification test (NAAT)
* Participants reporting receptive anal intercourse in the last 12 months: positive rectal gonorrhea or Chlamydia test by NAAT or culture
* Asthma other than mild, well-controlled asthma. More information on this criterion can be found in the protocol.
* History of partial or complete hysterectomy
* History of valvular heart disease
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Angioedema within the last 3 years if episodes are considered serious or have required medication within the last 2 years
* Hypertension. More information on this criterion can be found in the protocol.
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy. (Not excluded: a participant with a surgical excision and subsequent observation period that in the investigator's estimation has a reasonable assurance of sustained cure or is unlikely to recur during the period of the study.)
* Seizure disorder. (Not excluded: a participant with a history of seizures who has not required medications or had a seizure for 3 years.)
* Asplenia: any condition resulting in the absence of a functional spleen
* Psychiatric condition that precludes compliance with the protocol
* Pregnant or breastfeeding
* If born male, has been circumcised within 90 days prior to first vaccination or displays evidence that surgical site is not fully healed.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2011-05; Primary Completion 2013-09 (Actual); Study Completion 2017-11-22 (Actual)

PRIMARY OUTCOMES:
HIV-specific T-cell response rates detected in specimens collected from the rectum, semen, or cervix as assessed by IFN-γ ELISpot assay and/or flow cytometry | Throughout study

SECONDARY OUTCOMES:
Local and systemic reactogenicity signs and symptoms, adverse events and severe adverse events. | Throughout study
Induction of mucosal homing markers on HIV-specific T-cells as assessed by flow cytometric assays of peripheral blood samples | Throughout study
Multiparameter flow cytometric analyses of dendritic and NK cells in PBMCs, analysis of cytokines and chemokines using a multiplex assay of serum, plasma, semen, cervical secretions and dried blood spots, and gene expression analysis of RNA from PBMCs. | Throughout study
Flow cytometric analysis of T-cell activation and subsets detected in specimens collected from the rectum, semen, or cervix | Throughout study
Adenovirus-specific T-cell response rates detected in specimens collected from the rectum, semen, or cervix as assessed by IFN-γ ELISpot assay and/or flow cytometry | Throughout study
HIV-specific IgA and IgG responses in saliva, cervical secretions, semen, which may include neutralizing activity | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Janine Maenza, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Seattle Vaccine and Prevention CRS, Seattle, Washington, United States